CLINICAL TRIAL: NCT05470868
Title: Phase I Clinical Study, to Evaluate the Safety and Tolerability of the Ophthalmic Solution PRO-185 When Applied on the Ocular Surface of Healthy Volunteers
Brief Title: Safety and Tolerability of PRO-185
Acronym: PRO-185
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOPH185-0521/I
Record Dates: First submitted 2022-03-23; First posted 2022-07-22 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Hyperemia Eye
MeSH Terms: interventions — Naphazoline

STUDY DESIGN:
Intervention Model Description: Phase I, controlled, non-comparative, single-center, open study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRO-185 (Experimental): Healthy volunteers will apply one drop of PRO-185 ophthalmic solution (naphazoline / hypromellose) on both eyes, QID (four times per day) for 8 days.
  Interventions: Drug: Naphazoline / Hypromellose Ophthalmic

INTERVENTIONS:
Drug: Naphazoline / Hypromellose Ophthalmic — Naphazoline 0.03% / Hypromellose 0.2%

SUMMARY:
Phase I Study to evaluate safety and tolerability of PRO-185 (naphazoline/hypromellose) ophthalmic solution through evaluation of vital signs, ocular signs such as intraocular pressure, hyperemia and mydriasis and adverse events.

DETAILED DESCRIPTION:
A total of 22 healthy volunteers will apply PRO-185 ocular solution on both eyes QID (four times per day) for 8 days. The safety variables will include intraocular pressure, heart rate, systolic and diastolic blood pressure. Tolerability variables will include: hyperemia, mydriasis, and expected and unexpected adverse events. The presence of any of these in ≤ 20% will deem PRO-185 as safe and tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Being clinically healthy
* Having the ability to grant a signed informed consent
* Being able and willing to comply with the programmed visits, treatment plan and other procedures of this study.
* Age between 18 and 45 years
* Women in child-bearing age must assure the continuation (start ≥ 30 days previous to the signing of the ICF) of a hormonal contraceptive method or a intrauterine device (IUD) during the period of the study.
* Best corrected visual acuity equal of better than 20/30 in both eyes.
* Vital signs within normal ranges.
* Intraocular pressure ≥10 and ≤ 21 mmHg

Exclusion Criteria:

* Using any kind of topic ophthalmic products
* Presenting allergies to naphazoline or the history of intolerance to nasal decongestants or ocular vasoconstrictive products.
* History of diagnosis of suspicion of primary angle closure, primary angle closure or closed angle glaucoma.
* History of iridotomies or waiting for this procedure to take place.
* Conjunctival hyperemia grade 3 or 4 according to Efron scale.
* Ocular surface staining equal or greater to 3 in the SICCA scale, for any eye.
* Using medications or herbology products, through any route of administration.
* Pregnant, breastfeeding or women who plan to get pregnant during the period of the study.
* Previous participation in any clinical study 90 days prior to the inclusion in the present study.
* Previous participation in this study.
* Using contact lenses which cannot be suspended during the period of this study.
* History of any chronic illness, including diabetes and hypertension.
* Active inflammation or infection at the time of inclusion in this study.
* Unresolved lesions or traumas at the moment of inclusion in this study.
* History of any kind of ocular surgery.
* History of any surgical procedure, non-ophthalmologic, within the previous 3 months to the inclusion in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-02-04 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- IIMET Investigación e Innovación en Medicina Translacional, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PRO-185
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The manifested adverse events during the conduction of this trial were obtained during trial visits and reported in the electronic CRF, where the clinical team of the center included the information from source documents. These were previously checked by the monitor team, pharmacovigilance specialist, and the medical specialist part of the sponsor's crew to verify concordance with what was stipulated in the protocol.
Units Other Than Participants: Eyes
Arm/Group | PRO-185
Number analyzed (Participants) | 22
Number analyzed (Eyes) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.82 (4.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 22
Intraocular Pressure (IOP) [Mean (Standard Deviation); unit: mmhg] | 14.00 (2.80)
Pupillary diameter [Mean (Standard Deviation); unit: millimeters] | 6.50 (0.47)

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) Increment
Description: Safety evaluation through the incidence of subjects presenting an IOP elevation comparing Baseline Visit, Final Visit and before and after (20 minutes) research product administration (V1 and V2). Only right-eye values were analyzed.
Time Frame: Baseline visit (BV), day 1(pre and post pupil dilation); Visit 1 (V1), day 3 +1 (pre and post research product application); Visit 2 (V2), day 8 (pre and post research product application); Final Visit, day 10 (+1)
Measure: Mean (Standard Deviation); unit: mmhg
Units Other Than Participants: Eyes (right)
Arm/Group | PRO-185
Number analyzed (Participants) | 22
Number analyzed (Eyes (right)) | 22
mmhg
  VB IOP (pre-pupil dilation) | 14.00 (2.17)
  VB IOP (post-pupil dilation) | 13.57 (2.75)
  V1 IOP (pre-research product application) | 13.47 (2.21)
  V1 IOP (post-research product application) | 13.25 (1.90)
  V2 IOP (pre-research product application) | 13.02 (2.09)
  V2 IOP (post-research product application) | 13.65 (2.63)
  FV IOP | 12.79 (2.17)

2. Primary Outcome: Heart Rate Increment
Description: Safety evaluation through the incidence of subjects presenting an elevation > 15 beats per minute 20 minutes after administration, in comparison to baseline value.
Time Frame: Baseline visit, day 1(pre and post pupil dilation); Visit 1, day 3 +1 (pre and post research product application); Visit 2, day 8 (pre and post research product application); Final Visit, day 10 (+1)
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | PRO-185
Number analyzed (Participants) | 22
beats per minute
  BV Heart Rate | 73.27 (11.31)
  V1 Heart Rate (pre-instillation) | 70.54 (7.49)
  V1 Heart Rate (post70.59-instillation) | 70.59 (6.03)
  V2 Heart Rate (pre-instillation) | 70.68 (5.33)
  V2 Heart Rate (post-instillation) | 69.90 (4.61)
  FV Heart Rate | 73 (9.19)

3. Primary Outcome: Blood Pressure Increment (Systolic)
Description: Safety evaluation through the incidence of subjects presenting an elevation > 15 mmHg in systolic pressure or > 10 mmHg in diastolic pressure 20 minutes after administration, in comparison to baseline value.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PRO-185
Number analyzed (Participants) | 22
mmHg
  BV Systolic Blood Pressure | 113.81 (9.09)
  V1 Systolic Blood Pressure (pre-instillation) | 111.00 (12.07)
  V1 Systolic Blood Pressure (post-instillation) | 111.22 (10.72)
  V2 Systolic Blood Pressure (pre-instillation) | 107.50 (10.40)
  V2 Systolic Blood Pressure (post-instillation) | 108.63 (9.21)
  FV Systolic Blood Pressure | 113.90 (12.14)

4. Primary Outcome: Incidence of Conjunctival Hyperemia
Description: Tolerability evaluation through the incidence of conjunctival hyperemia grades 3 and 4 (according to the Efron scale). A higher score (grades) in this scale translates into worse outcomes. Only right-eye values were analyzed.
Time Frame: Trough Day 10 (+1)
Measure: Number; unit: Number of participants gde 3 or 4 Hypere
Units Other Than Participants: Eyes (right)
Arm/Group | PRO-185
Number analyzed (Participants) | 22
Number analyzed (Eyes (right)) | 22
Number of participants gde 3 or 4 Hypere | 2

5. Primary Outcome: Incidence of Pharmacological Mydriasis
Description: Incidence of pharmacological mydriasis measured through OPD III scan. If there was a change greater than 2 mm in pupil diameter between the baseline visit and any of the other measurements, pharmacological mydriasis was considered present, also if there was this change between the pre- and post-examination of the investigational product during visits 1 and 2.
Time Frame: Trough Day 10 (+1)
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes (right)
Arm/Group | PRO-185
Number analyzed (Participants) | 22
Number analyzed (Eyes (right)) | 22
millimeters | 6.50 (0.60)

6. Primary Outcome: Blood Pressure Increment (Diastolic)
Description: as for outcome 3
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PRO-185
Number analyzed (Participants) | 22
mmHg
  BV Diastolic Blood Pressure | 68.36 (8.16)
  V1 Diastolic Blood Pressure (pre-instillation) | 68.40 (7.73)
  V1 Diastolic Blood Pressure (post-instillation) | 69.45 (7.2)
  V2 Diastolic Blood Pressure (pre-instillation) | 66.59 (6.54)
  V2 Diastolic Blood Pressure (post-instillation) | 67.31 (7.67)
  FV Diastolic Blood Pressure | 67.41 (7.76)

ADVERSE EVENTS:
Time Frame: From day 1 (basal visit) to final visit on day 10 (±1 days)
Description: The manifested adverse events during the conduction of this trial were obtained during trial visits and reported in the electronic CRF, where the clinical team of the center included the information from source documents. These were previously checked by the monitor team, pharmacovigilance specialist, and the medical specialist part of the sponsor's crew to verify concordance with what was stipulated in the protocol.
Arm/Group | PRO-185
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 9/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRO-185 (N=22)
Burning sensation (Eye disorders) | 6
Headache (Nervous system disorders) | 1
Tearing (Eye disorders) | 2
Blurred vision (Eye disorders) | 1
Irritation in the area of instillation (Endocrine disorders) | 1
conjunctival hyperemia (Eye disorders) | 2
punctate keratitis (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT05470868/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05470868/SAP_001.pdf